CLINICAL TRIAL: NCT03426085
Title: The Effects of Liraglutide on Sudomotor Function and Inflammation in Type 2 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Aaron I. Vinik, MD, PhD, Professor of Medicine/Pathology/Neurobiology Director of Research & Neuroendocrine Unit, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-12-FB-0218
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Autonomic Nervous System Diseases; Sweat Gland Diseases; Diabetic Neuropathy With Neurologic Complication
MeSH Terms: conditions — Autonomic Nervous System Diseases; Sweat Gland Diseases; Diabetic Neuropathies | interventions — Liraglutide; Solutions; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Same formulation as active medication minus the active ingredient. Patients will start with 0.1 mL of liraglutide placebo and will escalate the dose every week in 0.1 ml increments until the 0.3 ml dose is reached. Escalation will be done according to patients' tolerance and glucose control
  Interventions: Other: Placebo
- Liraglutide 6 mg Solution for Injection (Experimental): After randomization, patients will undergo a treatment dose escalation phase. Liraglutide will be started at 0.6 mg SQ QD for 1 week, increased to 1.2 mg subcutaneous, per day (SQ, QD) for 1 week, and then increased and maintained on 1.8 mg SQ QD or maximally tolerated dose if self monitored blood glucose (SMBG) is at goal. Escalation will be done according to patients' tolerance and glucose control
  Interventions: Drug: Liraglutide 6 mg Solution for Injection

INTERVENTIONS:
Drug: Liraglutide 6 mg Solution for Injection
  Arms: Liraglutide 6 mg Solution for Injection
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to conduct an interventional, one year, randomized, double blind, placebo-controlled trial with Liraglutide in patients with type 2 diabetes (diabetes duration of >6 months and <10 years, HbA1c <10%) to evaluate its effects on the peripheral autonomic nervous system, as well as inflammatory markers, and measures of oxidative and nitrosative stress.

DETAILED DESCRIPTION:
The investigators propose to examine the effects of GLP-1 receptor agonist Liraglutide on autonomic sudomotor function and endothelial and neurovascular functions as well as markers of inflammation in patients with type 2 diabetes mellitus (T2DM). The primary objective will be changes in peripheral autonomic function using sudorimetry (Sudoscan) after 1 year of treatment.

The secondary objectives include changes on markers of inflammation and oxidative/nitrosative stress including C-reactive protein (CRP), interleukin 1 beta (IL-1β), Interleukin 6 (IL6), interleukin 12 (IL12), interleukin 10 (IL10), tumor necrosis factor α (TNF α), plasminogen activator Inhibitor 1 (PAI-1), superoxide dismutase (SOD), nitrotyrosine, carboxymethyl-lysine (CML), thiobarbituric acid reactive substances (TBARS), and asymmetric dimethylarginine (ADMA). Additional objectives include changes in neurovascular and endothelial function, measured by continuous Laser Doppler assessment of skin blood flow in response to different stimuli; and changes in sensory-motor peripheral nerve function, measured by clinical neuropathy scores (NSS & NIS), quantitative sensory testing and nerve conduction testing.

The aim of this study is to capture patients early in the disease process, when autonomic dysfunction is still potentially reversible. Several studies have shown the presence of autonomic imbalance in the early stages of diabetes and even in the pre-diabetic state (impaired glucose tolerance, impaired fasting glucose, and metabolic syndrome). We hypothesize that by treating type 2 diabetic patients with Liraglutide early in the disease process (<10 years of diagnosis), we will be able to improve peripheral autonomic imbalance, endothelial and neurovascular function, and reduce inflammation and oxidative/nitrosative stress. This will shed further insight into the mechanisms by which glucagon-like peptide-1 (GLP-1) exerts a neuroprotective role and improves the inflammatory process. The possibility of improving autonomic imbalance, endothelial function and inflammation may have important impact in the development of new potential therapeutic strategies to abrogate the microvascular complications of diabetes

ELIGIBILITY:
Inclusion Criteria:

1. established type 2 diabetes (diabetes duration of >6 months and <10 years).
2. Age 18-80 years
3. HbA1c at screening ≤ 10%
4. Subjects on stable (≥3 months prior to Screening) Standard of Care background diabetic therapy. Diabetic treatment regimens include diet and exercise alone or in association with oral anti-diabetic drugs (monotherapy or combinations) and/or long-acting insulin.

Exclusion Criteria:

1. Presence of type 1 diabetes mellitus (defined as C-peptide <1 ng /ml, <35y and prone to ketoacidosis)
2. Treatment with rapid-acting or short-acting insulin within the last 3 months
3. Proliferative retinopathy or maculopathy requiring acute treatment
4. Impaired renal function , defined as serum creatinine ≥ 125 µmol/L (≥1.4 mg/dL) for males and ≥ 110 µmol/L (≥1.24 mg/dL) for females
5. Impaired liver function, defined as aspartate transaminase (AST) or alanine transaminase (ALT), ≥ 2.5 times the upper limit of normal
6. Presence of clinically significant peripheral or autonomic neuropathy that is clearly of non-diabetic origin
7. Uncontrolled treated/untreated hypertension (systolic blood pressure (BP) ≥180 or diastolic blood pressure (BP) ≥100 at screening)
8. Clinically significant active macrovascular disease including myocardial infarction or cerebrovascular event within the past 6 months. Other exclusions include coronary artery bypass graft or coronary angioplasty in the previous 3 months, unstable angina pectoris (chest pain at rest, worsening chest pain, or admission to the emergency room (ER) or hospital for chest pain) within the previous 3 months, and/or congestive heart failure (NYHA Class III-IV)
9. Subjects known to be Hepatitis B surface antigen or Hepatitis C antibody positive with active hepatitis.
10. Active infection (e.g., human immunodeficiency virus (HIV), hepatitis), or a history of severe infection during the 30 days prior to screening
11. Evidence of immunocompromised status, including but not limited to individuals who have undergone organ transplantation, who are known to be HIV positive, or who are taking immunosuppressive drugs or chronic systemic corticosteroid treatment.
12. Major surgical procedure during the 30 days prior to screening
13. Diagnosis and/or treatment of malignancy (except for basal cell or squamous cell skin cancer, in-situ carcinoma of the cervix, or in-situ prostate cancer) within the past 5 years
14. Known clinically significant gastric emptying abnormality (e.g. severe gastroparesis), or history of gastric bypass (bariatric) surgery
15. Thyroid stimulating hormone (TSH) outside of normal limits at screening, or presence of a thyroid nodule detected on physical examination that has not been fully evaluated
16. Thyroid hormone therapy that has not been stable for ≥6 weeks prior to Screening
17. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN-2)
18. History of acute or chronic pancreatitis
19. Subjects taking medications that are known to affect autonomic function need to be at a stable dose of those medications ≥ 3 months prior to inclusion in the study
20. Other clinically significant, active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, genitourinary or hematological system that, in the opinion of the investigator, would compromise the subject's participation in the study, might confound the results of the study or pose additional risk in administering the study drug
21. Recurrent severe hypoglycemia and/or hypoglycemia unawareness.
22. Concurrent participation in another clinical trial with use of an experimental drug or device within 30 days of study entry.
23. Known or suspected history of alcohol or substance abuse
24. Mental incapacity, unwillingness or language barrier precluding adequate understanding of or cooperation with the study.
25. Women of childbearing potential (WOCBP*) who are pregnant, breast-feeding or intend to become pregnant
26. WOCBP* must have a negative pregnancy test at Screening and must agree to use adequate contraceptive methods** during the study and for one additional menstrual cycle following the end-of-treatment visit
27. Known or suspected hypersensitivity to study product(s) or related products
28. Patients with low vitamin B12 levels will be excluded
29. Current use or use 6 months prior to study participation of dipeptidyl peptidase-4 (DPP-4) inhibitors or glucagon like peptide-1 (GLP-1) agonists will be excluded
30. Liraglutide has not been studied in combination with prandial insulin. Patients who use prandial insulin may be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-04 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Sudomotor Function | One Year
  Changes in peripheral autonomic function using sudorimetry (Sudoscan) after 1 year of treatment.

SECONDARY OUTCOMES:
Inflammatory Markers C-Reactive Protein (CRP) | One year
  Changes on markers of inflammation and oxidative/nitrosative stress including C-reactive protein (CRP)
Inflammatory Markers IL-1β | One Year
  Changes on markers of inflammation and oxidative/nitrosative stress including IL-1β
Inflammatory Markers IL6 | One Year
  Changes on markers of inflammation and oxidative/nitrosative stress including IL6
Inflammatory Markers Tumor Necrosis factor α (TNF α) | One Year
  Changes on markers of inflammation and oxidative/nitrosative stress including Tumor Necrosis factor α (TNF α)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Vinik, MD, PhD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Strelitz Diabetes Center, Norfolk, Virginia, United States